CLINICAL TRIAL: NCT06867393
Title: Phase I Clinical Study of the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Oral Doses of HL-003 in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of HL-003 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HL-003-101
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subjects
Keywords: safety, tolerability; pharmacokinetic characteristics; HL-003 tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HL-003 tablet Placeco (Placebo Comparator)
  Interventions: Drug: HL-003 tablet Placeco
- HL-003 tablet (Active Comparator)
  Interventions: Drug: HL-003 tablet

INTERVENTIONS:
Drug: HL-003 tablet Placeco — 100mg、250mg、500mg、1000mg、1500mg，SAD
  Arms: HL-003 tablet Placeco
Drug: HL-003 tablet — 25mg、100mg、250mg、500mg、1000mg、1500mg，SAD
  Arms: HL-003 tablet

SUMMARY:
This clinical study aims to evaluate the safety, tolerability, and pharmacokinetic characteristics of HL-003 tablets in healthy subjects. It is conducted in two sequential clinical phases: single-dose and multiple-dose escalation.

DETAILED DESCRIPTION:
The single-dose escalation clinical trial of HL-003 tablets is designed as a dose-escalation, randomized, double-blind, placebo-controlled, parallel-group study.

The multiple-dose clinical trial of HL-003 tablets is designed as a randomized, double-blind, placebo-controlled, parallel-group study. The specific dosage, dosing frequency, and duration of continuous administration will be adjusted based on the results of the single-dose escalation clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers must be between 18 and 50 years old (inclusive), healthy, and can be of any gender.
2. Males must weigh ≥50 kg, and females must weigh ≥45 kg. The Body Mass Index (BMI) should be within the range of 19 to 26 kg/m² (including the threshold values).
3. Serum creatinine levels must be within the normal range during the screening period, and the Creatinine Clearance (CCr) must be ≥90 mL/min (including the threshold value, calculated using the CKD-EPI formula.
4. Comprehensive physical examination, vital signs, 12-lead electrocardiogram (ECG), chest X-ray (posteroanterior view), and laboratory tests (including blood routine, blood biochemistry, thyroid function, parathyroid function, coagulation function, urinalysis, etc.) must all be within normal ranges or show no clinically significant abnormalities.
5. Participants must agree not to plan for pregnancy during the trial and for 3 months after taking the medication, and must use reliable contraceptive methods.
6. Participants must be able to communicate effectively with researchers, fully understand the purpose, methods, requirements, and potential adverse reactions of the trial, voluntarily participate in the clinical trial, sign a written informed consent form, and be able to complete the clinical trial according to the protocol requirements.

Exclusion Criteria:

1. History of known allergy to the investigational drug or any of its components/related formulations; history of allergic reactions to two or more medications, foods, etc., or individuals with hypersensitive constitution;
2. Subjects with special dietary requirements who cannot comply with standardized meals;
3. History of frequent nausea or vomiting from any cause;
4. QTcF interval >450 msec (calculation formula in Appendix 14-3);
5. Positive for HBsAg, hepatitis B e-antigen, HCV antibody, syphilis antibody, or HIV antibody;
6. Consumption of caffeine-rich foods/beverages within 48h before dosing, or unwillingness to abstain during the study;
7. Any medical history/comorbidities that may affect safety assessment or drug metabolism, including CNS, cardiovascular, digestive, respiratory, urinary, hematologic, immunological, psychiatric disorders, metabolic abnormalities, or gastrointestinal surgery (except appendectomy);
8. Blood loss ≥400 mL or blood transfusion within 3 months before dosing; Blood donation (including component donation) ≥200 mL within 1 month before dosing;
9. Use of CYP3A4/CYP2C9/CYP2C8 inhibitors/inducers within 30 days before dosing; Any prescription/OTC medications/herbal products within 14 days before dosing;
10. Participation in other drug trials within 3 months before dosing;
11. Current/past drug addiction or positive drug abuse screening;
12. Excessive alcohol consumption (>14 units/week; 1 unit=360mL beer/45mL 40% liquor/150mL wine) within 3 months or unwillingness to abstain during the study;
13. Heavy smoking (>5 cigarettes/day within 3 months) or inability to abstain during the study;
14. Consumption of CYP-affecting foods (grapefruit/pomelo/lime products) within 48h before dosing, or refusal to abstain during the study;
15. Poor compliance or other investigator-determined unsuitable factors;
16. Additional female exclusions:

    1. Oral contraceptive use within 30 days before screening or during study
    2. Long-acting estrogen/progestin use within 6 months before screening
    3. Unprotected intercourse within 14 days before study or during trial
    4. Pregnancy or lactation;
17. Directly involved research staff or their family members, or subordinate researchers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-related adverse events (TRAEs) that were intolerable (requiring intervention) | up to 3 days
Incidence of TEAEs | up to 3 days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters: Tmax | up to 3 days
Pharmacokinetic (PK) parameters: Cmax | up to 3 days
Pharmacokinetic (PK) parameters: AUC0-t | up to 3 days
Pharmacokinetic (PK) parameters: AUC0-inf | up to 3 days
Pharmacokinetic (PK) parameters: t1/2 | up to 3 days
Pharmacokinetic (PK) parameters: CL/F | up to 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China